CLINICAL TRIAL: NCT00037050
Title: Linezolid vs. Vancomycin/Oxacillin/Dicloxacillin in the Treatment of Catheter-Related Gram-Positive Bloodstream Infections
Brief Title: Antibiotic Treatment for Infections of Short Term In-dwelling Vascular Catheters Due to Gram Positive Bacteria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M12600080; A5951060
Record Dates: First submitted 2002-05-14; First posted 2002-05-15 (Estimated); Last update posted 2009-09-14 (Estimated); Status verified 2009-09

CONDITIONS: Bacterial Infections; Gram-Positive Bacterial Infections; Bacteremia
MeSH Terms: conditions — Bacterial Infections; Gram-Positive Bacterial Infections; Bacteremia | interventions — Linezolid; Vancomycin; Oxacillin; Dicloxacillin

INTERVENTIONS:
Drug: Linezolid
  Other Names: Zyvox
Drug: Vancomycin
Drug: Oxacillin
Drug: Dicloxacillin

SUMMARY:
This study will treat patients who have a short term central catheter that is thought to be infected with a specific bacteria (gram positive bacteria)

ELIGIBILITY:
Inclusion Criteria:

* Patients with a central indwelling catheter with signs and symptoms of infection

Exclusion Criteria:

* Patients with tunneled catheter which cannot be removed.
* Patients with evidence of endovascular infection including endocarditis.
* Patients with infection of permanent intravascular devices.
* Patients who have received more than 1 day of another antibiotic before enrollment.
* Patients with HIV and low CD4 count.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 739 (Actual)
Dates: Start 2002-04; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The empiric treatment of patients with complicated skin and skin structure infections (cSSSI) related to an indwelling catheter;
The empiric treatment of patients with gram-positive catheter-related bloodstream infections.

SECONDARY OUTCOMES:
Clinical efficacy of linezolid compared to vancomycin/oxacillin/dicloxacillin.2.Incidence of late metastatic sequelae associated with S. aureus infections in patients treated with linezolid

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: Link to FDA Alert — http://www.fda.gov/Drugs/DrugSafety/PostmarketDrugSafetyInformationforPatientsandProviders/ucm101503.htm